CLINICAL TRIAL: NCT03831334
Title: An Open Label, Pilot Study Evaluating the Effect of Low-Dose Oral Minoxidil as Treatment of Permanent Chemotherapy-Induced Alopecia
Brief Title: Effect of Low-Dose Oral Minoxidil as Treatment of Permanent Chemotherapy-Induced Alopecia
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jennifer Nam Choi, MD, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JNC01142017
Record Dates: First submitted 2019-01-25; First posted 2019-02-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Permanent Chemotherapy-induced Alopecia
MeSH Terms: interventions — Minoxidil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Minoxidil Treatment (Experimental): Low dose oral minoxidil
  Interventions: Drug: oral minoxidil

INTERVENTIONS:
Drug: oral minoxidil — Participants will be provided with minoxidil (2.5 mg tablets) for 90 days (45 tablets + 5 extra in case of splitting difficulty) of treatment drug in dispensing containers and instructed to take half a pill (1.25mg), once a day.

SUMMARY:
An open label, pilot study involving the use of low dose oral minoxidil to treat permanent chemotherapy-induced alopecia.

DETAILED DESCRIPTION:
Patients will be evaluated through clinical assessment, histology, quality of life assessment, and adverse event monitoring. The data gathered from this study will be used to determine the safety and efficacy of the treatment regimen for this subset of CIA patients. The oral minoxidil regimen will be considered effective if significant clinical regrowth, positive histological changes, and improved Quality of Life are reported after the onset of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of permanent chemotherapy-induced alopecia who completed chemotherapy ≥ 6 months from the date of registration.
* Patients must be age ≥ 18 years.
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception (e.g., hormonal contraceptives such as birth control pills, patch, intrauterine device; barrier contraception such as male/female condoms, diaphragm; male partner with vasectomy; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of therapy.

Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

* FOCBP must have a negative urine or serum pregnancy test within 7 days prior to registration on study.
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration in the study.

Exclusion Criteria:

* Patients receiving any other investigational agents or using other alopecia treatments in the past 3 months are not eligible.
* Patients currently undergoing systemic cancer treatment or within 6 months of finishing chemotherapy are not eligible. Note: Patients receiving hormone modulators are eligible.
* Patients who have pheochromocytoma, hypothyroidism, anemia, cutaneous GVHD, hypotension, or a history of hypersensitivity to any components of the drug preparation are not eligible.
* Patients who have other forms of alopecia besides PCIA (with the exception of female pattern Ludwig 1 alopecia) are not eligible.
* Patients on oral or injectable anticoagulants are not eligible to participate in the optional punch biopsy
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible: (Uncontrolled Hypertension, Ongoing or active infection requiring systemic treatment, Symptomatic congestive heart failure, Unstable angina pectoris, Cardiac arrhythmia, Pericardial effusion, Psychiatric illness/social situations that would limit compliance with study requirements, Patients with any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints.)
* Patients currently taking guanethidine are not eligible. Patients may participate after a 1-week washout period.
* Patients currently taking drugs that may enhance the hypotensive effect of minoxidil are not eligible. Please contact study team regarding specific drug as washout period, as this will vary. Note: This includes: Alfuzosin, Amifostine, antipsychotic agents, Atazanavir, barbiturates, Benperidol, Brimonidine, Dapoxetine, Diazoxide, DULoxetine, Levodopa, Lormetazepam, Molsidomine, Naftopidil, Nicergoline, Nicorandil, Nitroprusside, Obinutuzumab, Pentoxifylline, phosphodiesterase 5 inhibitors, Probenecid, prostacyclin analogues, Quinagolide, and Valproate. If a patient is currently taking any of these drugs, further evaluation will be required to determine eligibility.
* Female patients who are pregnant or nursing are not eligible.
* Patients who have any condition or situation which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study are not eligible.
* Patients who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in degree of hair regrowth using the IPAQ scale | 48 weeks
  Evaluation will be performed by the investigators at each visit (every 12 weeks) as measured by the Investigator Photographic Assessment Questionnaire (IPAQ)
Change in degree of hair regrowth using the Dean Scale | 48 weeks
  Evaluation will be performed by the investigators at each visit (every 12 weeks) as measured by the Dean Scale

SECONDARY OUTCOMES:
Change in quality of life | 48 weeks
  Evaluation will be performed by the investigators at every other visit (every 24 weeks) until the end of the study (48 weeks total).The quality of life endpoint will be assessed with the Dermatology Life Quality Index (DLQI) as reported by the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Choi, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No